CLINICAL TRIAL: NCT02168478
Title: A Modified 48 Hour Patch Test of Neo-Synalar Cream, Sodium Lauryl Sulfate (Positive Control) and Saline (Negative Control)
Brief Title: Neo-Synalar Modified 48 Hour Patch Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Noah Rosenberg, MD (Industry)
Responsible Party: Sponsor-Investigator, Noah Rosenberg, MD, Chief Medical Officer, Medimetriks Pharmaceuticals, Inc
Organization: Medimetriks Pharmaceuticals, Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTWC01-001
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Allergy
Keywords: Neo-Synalar; Patch Test; Sodium lauryl sulfate; Saline; Presensitization
MeSH Terms: conditions — Hypersensitivity | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patch Test Group (Experimental): All subjects are patched with the following: 1.Neo-Synalar Cream 2.Sodium Lauryl Sulfate and 3. Saline.
  Test material is applied to the absorbent pad and allowed to remain in direct skin contact for a period of 48 hours.
  Interventions: Drug: Neo-Synalar Cream; Other: Sodium Lauryl Sulfate Aqueous Solution (0.40%); Other: Saline

INTERVENTIONS:
Drug: Neo-Synalar Cream — Approximately 0.2 g of test material is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Other Names: NS 0.5%(0.35% neomycin base)/ FA 0.025% Cream
Other: Sodium Lauryl Sulfate Aqueous Solution (0.40%) — Approximately 0.2 ml of the positive , 0.40% aqueous solution of sodium lauryl sulfate is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Other Names: SLS
Other: Saline — Saline is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.

SUMMARY:
A 48 hour patch test performed in healthy volunteers to determine the presensitization (pre-existing allergy) of Neo-Synalar (neomycin sulfate 0.5%(0.35% neomycin base), fluocinolone acetonide 0.025%) Cream . Subjects also receive a positive control (Sodium Lauryl Sulfate) and a negative control (Saline).

The primary objective of this study is to determine if any subjects exhibit an allergic reaction which may be indicative of a pre-existing sensitization.

DETAILED DESCRIPTION:
Following approximately 48 hours of continuous skin contact, the patch units and test material are removed at the testing facility. The test sites are evaluated for a significant reaction according to the ESS (Erythemal Scoring Scale).

The test sites are also re-evaluated at 96 and 168 hours post-application (for late reaction) using the ESS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 79 years inclusive.
* Subjects must be able to understand and execute informed consent.
* Female subjects must produce a negative pregnancy test.
* Subjects must be capable of following directions.
* Subjects must be considered reliable .

Exclusion Criteria:

* Subjects who are ill of health or taking medication that could influence the purpose, integrity, or outcome of the trial.
* Female subjects who are pregnant.
* Subjects with a history of adverse reactions to cosmetics, OTC (over the counter) drugs or other personal care products.
* Subjects who have used topical or systemic steroids or antihistamines within 7 days prior to trial initiation or plan to use either during the duration of the trial.
* Subjects with known allergy to neomycin, bacitracin, gentamicin, paromomycin, spectinomycin, streptomycin or tobramycin.
* Subjects with known allergy to corticosteroid.
* Subjects with a history of auto-immune disease (e.g. lupus, psoriatic arthritis, rheumatoid arthritis).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, Ph.D, Principal Investigator — Consumer Product Testing Corporation
Locations (1):
- Michael Caswell PhD., CCRC,CCRA, Fairfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited at single center- CPTC (Consumer Product Testing Corporation) located in Fairfield NJ.
Pre-assignment Details: There was no wash-out or run-in period
Groups:
- Patch Test Group: All subjects are patched with the following: 1.Neo-Synalar Cream 2.Sodium Lauryl Sulfate and 3. Saline.
  Test material is applied to the absorbent pad and allowed to remain in direct skin contact for a period of 48 hours.
  Neo-Synalar Cream: Approximately 0.2 g of test material is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Sodium Lauryl Sulfate Aqueous Solution (0.40%): Approximately 0.2 ml of the positive , 0.40% aqueous solution of sodium lauryl sulfate is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Saline: Saline is applied to the absorbent pad portion of a
Period: Overall Study
Arm/Group | Patch Test Group
Started | 206
Completed | 202
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Did Not Consent to Participation | 2
Not completed — Did Not Meet Exclusionary Criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Patch Test Group: All subjects are patched with the following: 1.Neo-Synalar Cream 2.Sodium Lauryl Sulfate and 3. Saline.
  All test material is applied to the absorbent pad and allowed to remain in direct skin contact for a period of 48 hours.
  Neo-Synalar Cream: Approximately 0.2 g of test material is applied to the absorbent pad portion of a semi-occlusive dressing and applied to upper back between the scapulae.
  Sodium Lauryl Sulfate Aqueous Solution (0.40%): Approximately 0.2 ml of the positive , 0.40% aqueous solution of sodium lauryl sulfate applied to the absorbent pad portion of a semi-occlusive dressing and applied to upper back between the scapulae.
  Saline: Saline is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae.
Arm/Group | Patch Test Group
Number analyzed (Participants) | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 170
  >=65 years | 31
Age, Continuous [Mean (Full Range); unit: years] | 48 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 202

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Pre-Existing Sensitization by Use of the Erythemal Scoring Scale (ESS)
Description: ESS is measured at 48, 96 and 168 hours post-application of study material. The Erythemal Scoring Scale (ESS) is defined as a 6 point scale (0-4). "0"= no visible erythema; "0.5"= slight, barely perceptible erythema; "1"= mild erythema; "2"= moderate erythema; "3"= marked erythema; "4"= severe erythema. An ESS score of 1 or greater that persists or worsens from one visit to the next is defined as pre-existing sensitization.
Time Frame: 48, 96 and 168 Hours
Measure: Number; unit: percentage of patients w allergic rxn
Groups:
- Patch Test Group: Neo-Synalar Cream: Approximately 0.2 g of test material is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Sodium Lauryl Sulfate Aqueous Solution (0.40%): Approximately 0.2 mL of the positive, 0.40% aqueous solution of sodium lauryl sulfate is applied to the absorbent pad portion of an occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
  Saline: Approximately 0.2 mL of saline is applied to the absorbent pad portion of an occlusive dressing and applied as received to the upper back between the scapulae. The patches are applied to a designated treatment site and allowed to remain in direct skin contact for a period of 48 hours.
Arm/Group | Patch Test Group
Number analyzed (Participants) | 202
percentage of patients w allergic rxn | 0

ADVERSE EVENTS:
Groups:
- Patch Test Group: All subjects are patched with the following: 1.Neo-Synalar Cream 2.Sodium Lauryl Sulfate and 3. Saline. Test material is applied to the absorbent pad and allowed to remain in direct skin contact for a period of 48 hours.
  Neo-Synalar Cream: Approximately 0.2 g of test material is applied to the absorbent pad portion of a semi-occlusive dressing and applied as received to the upper back between the scapulae.
  Sodium Lauryl Sulfate Aqueous Solution (0.40%): Approximately 0.2 ml of the positive , 0.40% aqueous solution of sodium lauryl sulfate is applied to the absorbent pad portion of an occlusive dressing and applied as received to the upper back between the scapulae.
  Saline: Approximately 0.2 ml of the saline is applied to the absorbent pad portion of an occlusive dressing and applied as received to the upper back between the scapulae.
Arm/Group | Patch Test Group
Serious Adverse Events (participants affected / at risk) | 0/202
Other Adverse Events (participants affected / at risk) | 0/202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No